CLINICAL TRIAL: NCT02854787
Title: Intravenous Bolus of Phenylephrine vs. Norepinephrine in Preventing Hypotension After Spinal Anesthesia for Cesarean Section
Brief Title: Intravenous Bolus of Phenylephrine vs. Norepinephrine in Preventing Hypotension After Spinal Anesthesia
Acronym: NorPN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, MD, assistant professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UniversityTunis el manar
Record Dates: First submitted 2016-07-30; First posted 2016-08-03 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-07

CONDITIONS: Anesthesia, Spinal and Epidural; Adverse Effect; Hypotension; Complications, Cesarean Section
Keywords: Spinal anesthesia; cesarean; blood pressure; Norepinephrine; Phenylephrine
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine (Active Comparator): A bolus of 100 mcg
  Interventions: Drug: Phenylephrine
- Norepinephrine (Active Comparator): A bolus of 0,2 mcg/kg
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — A bolus of 100 mcg
  Arms: Phenylephrine
Drug: Norepinephrine — A bolus of 0,2 mcg/kg
  Other Names: Noraline; Noradrénaline
  Arms: Norepinephrine

SUMMARY:
The purpose of the study is to determine if an intravenous bolus of phenylephrine is more effective compared to an intravenous bolus of norepinephrine associated with crystalloid loading for maintaining blood pressure during a spinal anesthetic for a cesarean delivery. Prevention of low blood pressure has been shown to decrease nausea and vomiting during and after cesarean delivery under spinal anesthesia. For elective cesarean delivery, all participants will receive spinal anesthesia with a local anesthetic and sufentanil. This study plans to enroll 120 pregnant women. Patients will be randomly assigned according to a computer generated system to be in one of two groups.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, active treatment controlled trial.

After written and informed consent are obtained, the study participants are randomly assigned using a computer generated table to 1 of 2 treatment groups prior to cesarean delivery.

Group A will consist of: An intravenous bolus of 0,2 mcg/Kg of norepinephrine to maintain systolic blood pressure (SBP) within 80-120% of baseline before the spinal.

Group B will consist of: An intravenous bolus of 100mcg of phenylephrine to maintain systolic blood pressure (SBP) within 80-120% of baseline before the spinal.

Patients will be admitted to holding area. Baseline arterial blood pressure and heart rate will be measured in supine position, with left uterine displacement. Baseline blood pressure will be calculated by taking the mean of three consecutive SBP measurements taken 5 minutes apart. 500 mL of Lactated Ringers solution will be administered immediately after induction of spinal anesthesia at the outflow rate of 100ml per hour.

The primary endpoint is the number of provider interventions needed to maintain the SBP within 100-120% of baseline for both groups. The secondary endpoint is nausea measured with each provider intervention after induction of spinal anesthesia, and immediately following delivery with 11 point verbal rating scale (0 = no nausea, 1 = nausea). Vomiting will be recorded whenever present during the surgical procedure.

Bradycardia (HR less than 50 BPM) will be treated with Atropine 0.4mg IV or ephedrine 3 mg - 12 mg IV bolus.

Study participants will receive a standard spinal anesthetic consisting of 0.5% hyperbaric bupivacaine (2 mL) plus sufentanil (5 mcg) at L3-4 or L4-5. Prior to surgical incision, the spinal sensory level will be tested to the bilateral T6-T4 dermatomal level. The patients will be positioned supine with a wedge placed under the right hip to avoid aortocaval compression. Both the patient and the researcher's assistant (who will collect data) will be blinded as to the administered Phenylephrine or norepinephrine bolus. The study will end when cesarean section is completed and the patient transferred to the post-operative care unit.

Measured variables will include systolic, diastolic and mean non-invasive blood pressure, the number and type of interventions for control of blood pressure, heart rate, incidence of nausea and vomiting (NV), incidence of arrhythmia and fetal cord blood analysis (pH) at delivery.

ELIGIBILITY:
Inclusion Criteria:

* of Anesthesiologists (ASA) Physical Status classification 1 and 2
* Pregnant women with singleton pregnancy

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maternal Blood Pressure | At time of surgery (right after spinal anesthesia until end of surgery)
  Measurement of systolic, diastolic and mean, non-invasive blood pressure during cesarean section with an infusion of either Ephedrine or Norepinephrine

SECONDARY OUTCOMES:
Hemodynamic Parameters - heart rate | At time of surgery (right after spinal anesthesia until end of surgery
  mean heart rate during cesarean section with an infusion of either Ephedrine or Norepinephrine
Hemodynamic Parameters - arrhythmia | At time of surgery (right after spinal anesthesia until end of surgery)
  incidence of arrhythmic events during cesarean section with an infusion of either Ephedrine or Norepinephrine
Vomiting | At time of surgery (right after spinal anesthesia until end of surgery)
  incidence of Vomiting (V) during cesarean section with an infusion of either Ephedrine or Norepinephrine. Measure will be done according to a simple scale: 0= no vomiting; 1= vomiting
mean pH of the fetal cord blood in each group | At time of birth
  fetal cord blood analysis will be done immediately after delivery in order to determine the pH value ( ie: logarithm of the blood concentration of hydrogen ions H+)in each group
Nausea | At time of surgery (right after spinal anesthesia until end of surgery)
  cesarean section with an infusion of either Ephedrine or Norepinephrine. Measure will be done according to a simple scale: 0= no nausea; 1= nausea

CONTACTS AND LOCATIONS:
Locations (1):
- Tunis maternity and neonatology center, minisetry of public health, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided